CLINICAL TRIAL: NCT07257289
Title: Stratification of Arrhythmic Risk and/or Heart Failure Risk in Patients With Hereditary Heart Disease
Acronym: PREVENT
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC25_0107
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sudden cardiac death (SCD) is one of the leading causes of death in developed countries. These deaths (more than 5,000 per year in France) are due to hereditary arrhythmias or cardiomyopathies. Early diagnosis of SCD is often achieved through family screening, but the main challenge is to stratify the risk of SCD in these patients. Indeed, prevention of SCD relies mainly on the implantation of an automatic defibrillator. The challenge is to identify patients who will develop SCD and avoid implanting an implantable cardioverter defibrillator (ICD) in patients who will never develop arrhythmias but who will face complications related to the ICD (inappropriate shocks, infection, lead failure), leading to a reduced quality of life and significant costs for the healthcare system. However, there is a lack of relevant clinical and biological markers for risk stratification, which rules out any possibility of preventive screening. Most of the clinical and ECG (electrocardiogram) parameters identifying an increased risk of SCD have not been reproduced in replication studies.

In this project, the investigator will develop a data processing and analysis pipeline using artificial intelligence methods to assess the individual risk of serious arrhythmic events or heart failure in patients with hereditary arrhythmic diseases or cardiomyopathies through the automated processing of multimodal data (clinical data, electrocardiogram (ECG), imaging (echocardiography, MRI magnetic resonance imaging), genetic data, biomarkers).

DETAILED DESCRIPTION:
The eligibility of patients (index cases and related cases) for the study will be determined during a cardiology consultation or day hospitalisation, carried out as part of routine care.

The investigator undertakes to obtain the person's free, informed and express consent, collected in writing, after providing them with oral and written information on the protocol and allowing them sufficient time to reflect. In the case of a minor patient, the investigator undertakes to inform the minor patient and their legal representatives orally and in writing and to obtain the minor's assent, i.e. their oral or written agreement depending on their age, and the written consent of their legal representatives.

Specific acts for research:

* Collection of two additional EDTA tubes (2 x 5 ml) during a blood test carried out as part of routine care, except for minors under the age of 4, for whom a saliva sample will be offered instead.
* Collection of one dry tube (5 ml) during a blood test carried out as part of routine care for biomarker analysis and only for adult patients.

Clinical data will be collected in a parameterised and secure eCRF (electronic Case Report Form).

Patients will be followed in the routine care for maximum 10 years. Arrhythmias, heart failure and sudden cardiac death will be collected during follow-up.

A data processing and analysis pipeline using artificial intelligence methods to assess the individual risk of serious arrhythmic events or heart failure in patients with hereditary arrhythmic diseases or cardiomyopathies through the automated processing of multimodal data (clinical data, electrocardiogram (ECG), imaging (echocardiography, MRI magnetic resonance imaging), genetic data, biomarkers) will be developped.

ELIGIBILITY:
Inclusion Criteria :

I. hereditary heart disease II. All relatives of patients III. Patients referred to the reference centre for suspected hereditary rhythm disorders or cardiomyopathies IV. Written consent V. social security scheme

Exclusion Criteria :

I. Patients participating in a therapeutic trial that may interfere with the research results II. Patients under guardianship or curatorship.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult and minor patients with hereditary heart disease or cardiomyopathies and their relatives.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2036-01-01 (Estimated); Study Completion 2036-12-12 (Estimated)

PRIMARY OUTCOMES:
Arrhythmic and heart failure risk stratification | 5, 8 and 10 years
  to assess the arrhythmic risk and/or risk of heart failure in patients with hereditary heart disease at 5, 8 and 10 years, using a model combining clinical, electrocardiographic, imaging, genetic and biomarker data.

SECONDARY OUTCOMES:
Demographics data | 5, 8 and 10 years
  Determine the risk of arrhythmia and/or heart failure based on demographics data
Diagnosis of Brugada syndrome | 5 years
  Evaluate the diagnostic performance of the model combining clinical, electrocardiographic, genetic and biomarker data for the identification of Brugada syndrome.

CONTACTS AND LOCATIONS:
Locations (15):
- France (13):
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CHU de La Rochelle, La Rochelle
  - CHU de Limoges, Limoges
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours
- CHU de la Martinique, Fort-de-France, Martinique
- CHU de la Réunion, Saint-Pierre, Reunion